CLINICAL TRIAL: NCT06403787
Title: Effect of Implementing an Aerobic Training Program and Administering Ginkgo Biloba Extract on Plasma Concentrations of LDL and HDL in HIV Positive Patients Undergoing Antiretroviral Treatment at the HIV Unit of Hospital Civil Fray Antonio Alcalde
Brief Title: Effect of Aerobic Training and Ginkgo Biloba on Lipids Levels in HIV-positive Patients Undergoing Antiretroviral Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Raul Soria Rodriguez, PhD, Associate Research Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-02922
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV-positive individuals; Aerobic exercise training; Ginkgo biloba extract; Plasma lipid concentrations
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Exercise; Ginkgo biloba extract; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Double-blind clinical trial with random allocation into three groups, all undergoing aerobic training. One group will receive ginkgo biloba extract, another will be administered atorvastatin, and a third will receive a placebo of calcined magnesia
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ginkgo biloba group (Experimental): This group will assess the effects of aerobic exercise combined with ginkgo biloba extract
  Interventions: Drug: Aerobic exercise + Ginkgo Biloba Extract
- Placebo group (Placebo Comparator): Participants in this group will serve as a control to evaluate the effects of aerobic exercise when administered a placebo of calcined magnesia
  Interventions: Drug: Aerobic exercise + Calcined magnesia (placebo)
- Statins group (Active Comparator): In this group, the effects of aerobic exercise along with the administration of atorvastatin will be investigated
  Interventions: Drug: Aerobic exercise + Atorvastatin

INTERVENTIONS:
Drug: Aerobic exercise + Ginkgo Biloba Extract — 12 weeks of intervention for the participants, divided into 3 stages implementing an exercise adaptation period. The adaptation period will span the first 4 weeks of the intervention, during which participants will be brought to an intensity between 50% and 60% of their maximum heart rate (HRmax). From week 5 to 8, the HRmax range will be increased from 60% to 70%, and during the last 4 weeks, it will be maintained at 70% of HRmax combined with 240 mg of LIFE EXTENSION® brand ginkgo biloba extract in 120 mg tablets
  Arms: Ginkgo biloba group
Drug: Aerobic exercise + Calcined magnesia (placebo) — 12 weeks of intervention for the participants, divided into 3 stages implementing an exercise adaptation period. The adaptation period will span the first 4 weeks of the intervention, during which participants will be brought to an intensity between 50% and 60% of their maximum heart rate (HRmax). From week 5 to 8, the HRmax range will be increased from 60% to 70%, and during the last 4 weeks, it will be maintained at 70% of HRmax combined with calcined magnesia (homogenized to the same weight of ginkgo biloba)
  Arms: Placebo group
Drug: Aerobic exercise + Atorvastatin — 12 weeks of intervention for the participants, divided into 3 stages implementing an exercise adaptation period. The adaptation period will span the first 4 weeks of the intervention, during which participants will be brought to an intensity between 50% and 60% of their maximum heart rate (HRmax). From week 5 to 8, the HRmax range will be increased from 60% to 70%, and during the last 4 weeks, it will be maintained at 70% of HRmax combined with 20 mg of atorvastatin
  Arms: Statins group

SUMMARY:
The administration of antiretroviral drugs (ART) has significantly prolonged the life expectancy of people living with human immunodeficiency virus (HIV) and delayed the progression towards Acquired Immune Deficiency Syndrome (AIDS). However, this has led to the emergence of other conditions, such as dyslipidemia, among individuals undergoing ART. Dyslipidemia is commonly managed with statin therapy, which has not been reported to have pharmacological interactions with ART. Additionally, ginkgo biloba extract (GBS) has been observed to improve blood lipid concentrations, and aerobic exercise training (EXA) interventions have shown positive modifications in these values.

Given this context, the present study aims to investigate the potential positive effects of an aerobic training program and the consumption of ginkgo biloba extract on plasma lipid concentrations in HIV-positive individuals. The study seeks to provide insights into novel strategies for managing dyslipidemia in this population.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 60 years
* Diagnosis of HIV-1 infection
* Receiving antiretroviral therapy with a triple regimen (Biktarvy treatment)
* Undetectable viral load (< 20 copies/mL) for the past 6 months CD4+ level > 200 cells/μL
* Diagnosis of mixed dyslipidemia in the last three months, indicated by:

  * Total cholesterol ≥ 200 mg/dL
  * HDL cholesterol < 40 mg/dL in men and < 50 mg/dL in women
  * LDL cholesterol > 100 mg/dL
* Triglycerides ≥ 150 mg/dL
* Possession of a mobile device or computer with internet access and necessary platforms
* Willingness to participate voluntarily in the study and provide written consent

Exclusion Criteria:

* Individuals who develop hypersensitivity or allergy to ginkgo biloba extract
* Failure to attend at least 80% of the physical exercise sessions (equivalent to missing more than 12 sessions)
* Lack of adherence to pharmacological treatment
* Participant's decision to discontinue the intervention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Comparison of changes in serum lipid levels. | 12 weeks
  Levels of Total Cholesterol (mg/dL), HDL (High-Density Lipoprotein) (mg/dL), LDL (Low-Density Lipoprotein) (mg/dL), VLDL (Very Low-Density Lipoprotein) (mg/dL) and, Triglycerides (mg/dL) will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Raul Soria Rodriguez, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- University Center for Health Sciences, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No